CLINICAL TRIAL: NCT01473849
Title: Non-interventional, Prospective Study to Evaluate the Impact of CMV Replication Over Hepatitis C Recurrence in Liver Transplant Recipients
Brief Title: Impact of Cytomegalovirus (CMV) Replication Over Hepatitis C Recurrence in Liver Transplant Recipients
Acronym: VHENUS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sociedad Española de Trasplante Hepático (Network)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Dr. Manuel de la Mata García, Sociedad Española de Transplante Hepático
Other Study IDs: VHENUS
Record Dates: First submitted 2011-05-30; First posted 2011-11-17 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Cytomegalovirus Infection; Hepatitis C
Keywords: Cytomegalovirus; Liver transplantation; Hepatitis C virus; Patients who underwent first liver transplantation due to hepatopathy caused by HCV,confirmed by detection of HCV RNA previously to transplantation
MeSH Terms: conditions — Cytomegalovirus Infections; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The relationship between cytomegalovirus infection and recurrence of hepatitis C in liver transplant recipients remains controversial. Although some studies (Teixeira et al., 2000; Singh et al., 2005)have not found an association between recurrence of hepatitis C and CMV infection, studies such as Rosen et al. show that 50% of patients with CMV infection suffered cirrhosis durig follow-up period, while between not-infected patients the rate was 11%. To clarify this question, a non-interventional study will be carried out in order to assess if CMV replication is a risk factor for graft dysfunction in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who underwent liver transplantation after hepatopathy caused by HCV, confirmed by pre-transplantation detection of HCV RNA
* Age > 18 years old

Exclusion Criteria:

* Patients co-infected with HBV or HIV
* Patients who show other causes of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver transplantation after hepatopathy caused by HCV
Sampling Method: Non-Probability Sample
Enrollment: 179 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Effect of CMV replication over hepatitis C recurrence | 48 weeks after transplantation
  viral charge of HCV will be assessed 48 weeks after transplantation

SECONDARY OUTCOMES:
Effect of CMV replication over fibrosis in graft after Hepatitis C recurrence after transplantation | 1 year
Effect of CMV recurrence over graft and patient survival | 1 year
Relationship between viral charge of CMV and HCV during study period | 1 year

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Carlos Haya, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza